CLINICAL TRIAL: NCT00424463
Title: An Expanded Controlled Study of MCI-186 for Treatment of Amyotrophic Lateral Sclerosis in Double-Blind, Parallel-Group, Placebo-Controlled Manner (Phase 3)
Brief Title: Expanded Controlled Study of Safety and Efficacy of MCI-186 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI186-17
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic lateral sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: MCI-186
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo of MCI-186

INTERVENTIONS:
Drug: MCI-186 — Two ampoules (60 mg) of MCI-186 injection are intravenously administered once a day for 10 days during 14 days, followed by 14 days observation period (first cycle). Then treatment (10 days' administration during 14 days ) - observation (14 days) cycle is repeated eight times.
  Other Names: Edaravone; Radicut
  Arms: 1
Drug: Placebo of MCI-186 — Two ampoules of placebo injection are intravenously administered once a day for 10 days during 14 days, followed by 14 days observation period (first cycle). Then treatment (10 days' administration during 14 days) - observation (14 days) cycle is repeated eight times.
  Arms: 2

SUMMARY:
This is a long-term, double-blind, placebo-controlled study of MCI-186 to treat ALS. This study is the long-term extension of Study NCT00330681; Study NCT00330681 is a Phase 3, randomized, double-blind, placebo control, parallel assignment, 24-week study in the treatment of ALS. The objectives of this study are to assess the efficacy and safety of long-term intermittent therapy with 60 mg MCI-186 to ALS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who ware completed drug administration without discontinuation in the preceding confirmatory study NCT00330681.

Exclusion Criteria:

* Patients with such complications as Parkinson's disease, schizophrenia, dementia, renal failure, or other severe complication, and patients who have the anamnesis of hypersensitivity to edaravone.
* Patients whose creatinine clearance is 50mL/min or less at the time of completion of drug administration in the study NCT00330681.
* Pregnant, lactating, and probably pregnant patients, and patients who want to become pregnant, and patients who can not agree to contraception.
* Patients who are participating in other clinical trials except the study NCT00330681.
* In addition to the above exclusion criteria, patients judged to be inadequate to participate in this study by their physician.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2007-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koji Abe, professor, Study Chair — Graduate School of Medicine and Dentistry, Okayama University
Locations (1):
- National Hospital Organization Miyagi National Hospital, Watari-gun, Miyagi, Japan

REFERENCES:
- [Result] WRITING GROUP ON BEHALF OF THE EDARAVONE (MCI-186) ALS 17 STUDY GROUP. Exploratory double-blind, parallel-group, placebo-controlled extension study of edaravone (MCI-186) in amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2017 Oct;18(sup1):20-31. doi: 10.1080/21678421.2017.1362000. PMID 28872918
- [Derived] Takahashi F, Takei K, Tsuda K, Palumbo J. Post-hoc analysis of MCI186-17, the extension study to MCI186-16, the confirmatory double-blind, parallel-group, placebo-controlled study of edaravone in amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2017 Oct;18(sup1):32-39. doi: 10.1080/21678421.2017.1361442. PMID 28872914

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-186 - Placebo of MCI-186: Cycles 7 to 12 (6 cycles) : 2 ampoules of edaravone injection placebo administered once daily over 60 minutes by intravenous infusion Cycles 13 to 15 (3 cycles) : 2 ampoules of edaravone injection 30 mg administered once daily over 60 minutes by intravenous infusion
- MCI-186 - MCI-186; Placebo of MCI-186 - MCI-186: Cycles 7 to 12 (6 cycles) : 2 ampoules of edaravone injection 30 mg administered once daily over 60 minutes by intravenous infusion Cycles 13 to 15 (3 cycles) : 2 ampoules of edaravone injection 30 mg administered once daily over 60 minutes by intravenous infusion
Period: Overall Study
Arm/Group | MCI-186 - Placebo of MCI-186 | MCI-186 - MCI-186 | Placebo of MCI-186 - MCI-186
Started | 45 | 48 | 88
Completed | 38 | 34 | 72
Not Completed | 7 | 14 | 16
Not completed — Adverse Event | 2 | 3 | 2
Not completed — Physician Decision | 0 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 2 | 5
Not completed — Tracheotomy due to worsening of ALS | 1 | 7 | 6
Not completed — Patient's convenience | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI-186 - Placebo of MCI-186 | MCI-186 - MCI-186 | Placebo of MCI-186 - MCI-186 | Total
Number analyzed (Participants) | 45 | 48 | 88 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 29 | 62 | 129
  >=65 years | 7 | 19 | 26 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 22 | 31 | 65
  Male | 33 | 26 | 57 | 116

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Revised ALS Functional Rating Scale (ALSFRS-R) Score in Full Analysis Set (FAS) Population at 24 Weeks
Description: 0=worst; 48=best To investigate the sustainability of effects of edaravone, the analysis focusing on the comparison between the placebo and edaravone groups of patients who had received 6 cycles of edaravone treatment, i.e., the comparison of data from Cycles 7 to 12 between the edaravone-edaravone group and the edaravone-placebo group, was performed.
Time Frame: baseline (seventh cycle) and at 24 week (twelfth cycle)
Population: "1 patient with diseases other than ALS" and "4 patients with missing data" were excluded from the FAS in the MCI-186 - Placebo of MCI-186group.
  "5 patients with missing data" were excluded from the FAS in the MCI-186 - MCI-186 group.
  "14 patients with missing data" were excluded from the FAS in the Placebo of MCI-186 - MCI-186 group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI-186 - Placebo of MCI-186 | MCI-186 - MCI-186 | Placebo of MCI-186 - MCI-186
Number analyzed (Participants) | 40 | 43 | 74
units on a scale | -5.5 (4.6) | -4.2 (4) | -5.4 (4.5)

2. Secondary Outcome: Number of Participants With Death or a Specified State of Disease Progression
Description: Any of "death, disability of independent ambulation, loss of upper arm function, tracheotomy, use of respirator, and use of tube feeding" was defined as an event.
Time Frame: 24 weeks (from seventh cycle to twelfth cycle)
Population: "1 patient with diseases other than ALS" was excluded from the FAS in the MCI-186 - Placebo of MCI-186 group.
Measure: Count of Participants; unit: Participants
Arm/Group | MCI-186 - Placebo of MCI-186 | MCI-186 - MCI-186 | Placebo of MCI-186 - MCI-186
Number analyzed (Participants) | 44 | 48 | 88
Participants
  death | 1 | 1 | 1
  disability of independent ambulation | 8 | 11 | 20
  loss of upper arm function | 3 | 5 | 7
  tracheotomy | 0 | 0 | 2
  use of respirator | 0 | 1 | 2
  use of tube feeding | 1 | 1 | 8

3. Secondary Outcome: Change From Baseline in % Forced Vital Capacity (%FVC) in Full Analysis Set (FAS) Population at 24 Weeks
Description: To investigate the sustainability of effects of edaravone, the analysis focusing on the comparison between the placebo and edaravone groups of patients who had received 6 cycles of edaravone treatment, i.e., the comparison of data from Cycles 7 to 12 between the edaravone-edaravone group and the edaravone-placebo group, was performed.
Time Frame: baseline (seventh cycle) and at 24 week (twelfth cycle)
Population: "1 patient with diseases other than ALS" and "4 patients with missing data" were excluded from the FAS in the MCI-186 - Placebo of MCI-186group.
  "6 patients with missing data" were excluded from the FAS in the MCI-186 - MCI-186 group.
  "19 patients with missing data" were excluded from the FAS in the Placebo of MCI-186 - MCI-186 group.
Measure: Mean (Standard Deviation); unit: percentage of FVC
Arm/Group | MCI-186 - Placebo of MCI-186 | MCI-186 - MCI-186 | Placebo of MCI-186 - MCI-186
Number analyzed (Participants) | 40 | 42 | 69
percentage of FVC | -10.6 (13.16) | -12.91 (14.97) | -10.54 (13.21)

4. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: 36 weeks (from seventh cycle to fifteenth cycle)
Measure: Number; unit: percentage of participant
Arm/Group | MCI-186 - Placebo of MCI-186 | MCI-186 - MCI-186 | Placebo of MCI-186 - MCI-186
Number analyzed (Participants) | 45 | 48 | 88
percentage of participant | 97.8 | 91.7 | 92

5. Secondary Outcome: Percentage of Participants With Adverse Drug Reactions
Time Frame: 36 weeks (from seventh cycle to fifteenth cycle)
Measure: Number; unit: percentage of participant
Arm/Group | MCI-186 - Placebo of MCI-186 | MCI-186 - MCI-186 | Placebo of MCI-186 - MCI-186
Number analyzed (Participants) | 45 | 48 | 88
percentage of participant | 4.4 | 10.4 | 10.2

6. Secondary Outcome: Percentage of Participants With Laboratory Tests for Which the Incidence of Abnormal Changes Was 5% or Higher in Either Group
Time Frame: 36 weeks (from seventh cycle to fifteenth cycle)
Measure: Number; unit: percentage of participant
Arm/Group | MCI-186 - Placebo of MCI-186 | MCI-186 - MCI-186 | Placebo of MCI-186 - MCI-186
Number analyzed (Participants) | 45 | 48 | 88
percentage of participant
  White blood cell count | 11.1 | 4.2 | 10.2
  Alanine aminotransferase | 0 | 6.3 | 4.5
  Urinary glucose | 0 | 6.3 | 3.4

7. Secondary Outcome: Percentage of Participants With Abnormal Changes in Sensory Examinations
Time Frame: 36 weeks (from seventh cycle to fifteenth cycle)
Measure: Number; unit: percentage of participant
Arm/Group | MCI-186 - Placebo of MCI-186 | MCI-186 - MCI-186 | Placebo of MCI-186 - MCI-186
Number analyzed (Participants) | 45 | 48 | 88
percentage of participant
  Numbness | 0 | 0 | 0
  Staggering | 0 | 2.1 | 2.3
  Vibratory sensation | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: from baseline (seventh cycle) to 36 weeks (fifteenth cycle)
Arm/Group | MCI-186 - Placebo of MCI-186 | MCI-186 - MCI-186 | Placebo of MCI-186 - MCI-186
Serious Adverse Events (participants affected / at risk) | 13/45 | 25/48 | 39/88
Other Adverse Events (participants affected / at risk) | 43/45 | 43/48 | 74/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-186 - Placebo of MCI-186 (N=45) | MCI-186 - MCI-186 (N=48) | Placebo of MCI-186 - MCI-186 (N=88)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 6 | 9 | 22
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abasia (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 0 | 4 | 5
Bronchitis (Infections and infestations) | 1 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 4 | 6 | 10
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Dyslalia (Nervous system disorders) | 1 | 0 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 6
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-186 - Placebo of MCI-186 (N=45) | MCI-186 - MCI-186 (N=48) | Placebo of MCI-186 - MCI-186 (N=88)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 2
Cataract (Eye disorders) | 1 | 2 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 3
Conjunctivitis allergic (Eye disorders) | 2 | 1 | 0
Dry eye (Eye disorders) | 1 | 1 | 1
Eye discharge (Eye disorders) | 0 | 0 | 2
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 8 | 10 | 20
Dental caries (Gastrointestinal disorders) | 0 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 6
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 2 | 2
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0 | 1
Malocclusion (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 3
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 0 | 2
Stomach discomfort (Gastrointestinal disorders) | 2 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 4
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 2
Catheter site erythema (General disorders) | 0 | 2 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 1
Feeling abnormal (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 9 | 10 | 27
Impaired healing (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 3 | 2
Thirst (General disorders) | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 3
Seasonal allergy (Immune system disorders) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 2 | 0 | 3
Catheter site infection (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0
Enterocolitis viral (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 1
Infected epidermal cyst (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 12 | 10 | 28
Oral herpes (Infections and infestations) | 0 | 1 | 2
Otitis media (Infections and infestations) | 0 | 1 | 0
Periodontal infection (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 2
Sinobronchitis (Infections and infestations) | 1 | 0 | 0
Sweat gland infection (Infections and infestations) | 0 | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 1 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 3 | 3 | 4
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Avulsion fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 7 | 3 | 8
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 1 | 2
Post gastric surgery syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 3
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2
Blood potassium increased (Investigations) | 0 | 1 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1
Glucose urine present (Investigations) | 0 | 1 | 2
White blood cell count increased (Investigations) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 4
Hyposmia (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 2 | 0 | 3
Insomnia (Psychiatric disorders) | 3 | 5 | 7
Dysuria (Renal and urinary disorders) | 0 | 0 | 2
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 3 | 3 | 3
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 2
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 8
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other